CLINICAL TRIAL: NCT05793060
Title: Dexmedetomidine Versus Dexamethasone as Adjuvants to Bupivacaine for Ultrasound-guided Intermediate Cervical Plexus Block in Patients Undergoing Thyroidectomy
Brief Title: Dexmedetomidine Versus Dexamethasone as Adjuvants to Bupivacaine for Intermediate Cervical Plexus Block
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Damanhour Teaching Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DTH: 23001
Record Dates: First submitted 2023-03-17; First posted 2023-03-31 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-07

CONDITIONS: Analgesia
Keywords: Cervical plexus block; Dexamethasone; Dexmedetomidine; Thyroidectomy
MeSH Terms: conditions — Agnosia | interventions — Dexmedetomidine; dexamethasone 21-phosphate; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (n=30) (Active Comparator): Dexmedetomidine group
  Interventions: Drug: Dexmedetomidine Hydrochloride
- Group B (n=30) (Active Comparator): Dexamethasone group
  Interventions: Drug: Dexamethasone Phosphate

INTERVENTIONS:
Drug: Dexmedetomidine Hydrochloride — Dexmedetomidine 50 Mcg
  Other Names: Precedex
  Arms: Group A (n=30)
Drug: Dexamethasone Phosphate — Dexamethasone 4 mg
  Other Names: Dexamethasone
  Arms: Group B (n=30)

SUMMARY:
Background: Many thyroidectomy patients suffer from postoperative pain that could delay early hospital discharge and place a significant burden on both the patient and the healthcare team. Bilateral intermediate cervical plexus block (ICPB) provides good analgesia for neck surgery, including thyroidectomy. However, the duration of a single-shot nerve block is usually short. Therefore, adjuvants are used in peripheral nerve blocks.

Objectives: To compare the safety and efficacy of dexmedetomidine versus dexamethasone as adjuvants to bupivacaine in ultrasound-guided intermediate cervical plexus block in patients undergoing total thyroidectomy under general anesthesia.

Patients and Methods: This is a randomized, double-blind, phase four, prospective clinical trial; carried out on 60 patients, who were candidates for total thyroidectomy under general anesthesia at our hospital. Patients were randomly allocated into two equal groups; group A, received bilateral ICPB with isobaric bupivacaine plus dexmedetomidine, and group B, received bilateral ICPB with isobaric bupivacaine plus dexamethasone.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status ≤ II
* Age from 21 to 60 years
* Body Mass Index (BMI) ≤ 35 kg/m2

Exclusion Criteria:

* ASA physical status > II
* Age < 21 years or > 50 years
* BMI > 35 kg/m2
* Bronchial asthma
* Chronic obstructive pulmonary disease
* Restrictive lung diseases
* Sick sinus syndrome
* Sinus bradycardia
* Hypertension
* Chronic hypotension
* Ischemic heart disease
* Coagulopathies
* Hepatic insufficiency
* Renal insufficiency
* Diabetes mellitus
* Peripheral neuropathy
* Thyroid malignancy
* Hyperthyroidism
* Substernal goiter
* Patients on beta-blockers
* Patients using pacemakers
* Alcohol or drug abuse
* Allergy to the study drugs

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Median and Range of Numeric Pain Rating Scale (NPRS) score [(median (range)] | 24 hours after the end of the operation
  NPRS measures the severity of pain, it is a 11 point scale from 0-10; where 0=No pain and 10=Worst possible pain ( At post anesthesia care unit (PACU), then every 2 hours till 24 hours)
Mean and Standard deviation of Numeric Pain Rating Scale (NPRS) score (mean±SD) | 24 hours after the end of the operation
  NPRS measures the severity of pain, it is a 11 point scale from 0-10; where 0=No pain and 10=Worst possible pain ( At PACU, then every 2 hours till 24 hours)

SECONDARY OUTCOMES:
Number of participants and Percentage of Drug-related side effects | 24 hours after the end of the operation
  Number of participants and Rate of: Bradycardia, Hypotension, Dysrhythmia, and Postoperative nausea and vomiting (PONV)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Shaat, MD, Principal Investigator — Damanhour Teaching Hospital
Locations (1):
- Damanhour Teaching Hospital, Damanhūr, El-Beheira, Egypt